CLINICAL TRIAL: NCT01079793
Title: A Phase I/II Study of Adjuvant Prostate Irradiation and Ixabepilone For High Risk Prostate Cancer Post-Prostatectomy
Brief Title: Radiation Therapy and Ixabepilone in Treating Patients With High-Risk Stage III Prostate Cancer After Surgery
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Overlapping study, PI preferred to enroll in alternate trial.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-09809; CDR0000666842 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ixabepilone; Chemotherapy, Adjuvant; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ixabepilone (Experimental): Adjuvant therapy
  Interventions: Drug: ixabepilone; Procedure: adjuvant therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: ixabepilone
Procedure: adjuvant therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Ixabepilone may also make tumor cells more sensitive to radiation therapy. Giving radiation therapy with chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ixabepilone when given together with radiation therapy to see how well it works in treating patients with high-risk stage III prostate cancer after surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose and dose-limiting toxicity of ixabepilone in combination with concurrent intensity-modulated radiation therapy in patients with high-risk prostate cancer after prostatectomy. (Phase I)
* To determine the toxicity profile of this regimen in these patients. (Phase I)

Secondary

* To assess freedom from progression in patients treated with this regimen. (Phase II)
* To assess biochemical failure, local failure, and distant failure in patients treated with this regimen. (Phase II)
* To assess disease-specific survival and overall survival of patients treated with this regimen. (Phase II)
* To evaluate acute and late toxicity of this regimen in these patients.

OUTLINE: This is a phase I, dose-escalation study of ixabepilone followed by a phase II study.

Patients undergo adjuvant intensity-modulated radiation therapy once daily, 5 days a week, for 7-9 weeks. Patients also receive concurrent ixabepilone IV over 1 hour on days 1 and 8. Treatment with ixabepilone repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 3 years, and then annually for 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Must have undergone any common form of prostatectomy (e.g., open, perineal, laparoscopic, or robotic) within the past 2 years
  * T3 disease or positive surgical margins
  * Node negative (N0) and free of distant metastasis (M0) by a bone scan and CT scan or MRI of the pelvis within the past 90 days
  * Considered high-risk disease
* Gleason score = 7 and post-operative PSA > 0 and ≤ 2 ng/mL OR Gleason score ≥ 8 and post-operative PSA ≥ 0 and ≤ 2 ng/mL
* Pre-prostatectomy PSA available

  * Range of pre-prostatectomy PSA values not required

PATIENT CHARACTERISTICS:

* Zubrod (ECOG) performance status 0-1
* ANC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN
* Fertile patients must use effective contraception during and for 4 weeks after completion of study therapy
* Patients with urinary incontinence waiting for stabilization of urinary function after prostatectomy allowed for up to 6 months
* No CTCv4 peripheral neuropathy (motor or sensory) ≥ grade 1
* No history of inflammatory colitis including Crohn disease or ulcerative colitis
* No significant history of psychiatric illness
* No other invasive malignancy within the past 3 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the oral cavity
* No severe, active co-morbidity with any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days
  * Immunocompromised patients or AIDS based upon current CDC definition

    * HIV testing not required
* No history of hypersensitivity reactions to agents containing Cremophor® EL or its derivatives (e.g., polyoxyethylated castor oil)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic radiotherapy or radiotherapy for another malignancy that encompasses ≥ 30% of major bone marrow-containing areas (e.g., pelvis or lumbar spine)
* No prior hormonal therapy for prostate cancer

  * Prior hormonal agents, e.g., finasteride or dutasteride, for benign prostatic hypertrophy allowed
* No other concurrent adjuvant antineoplastic therapy planned while on this protocol, including the following:

  * Cryotherapy
  * Hormonal therapy
  * Other chemotherapy for prostate cancer

    * Prior chemotherapy for a different type of cancer allowed provided it was administered > 3 years ago

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2011-10-17 (Actual); Study Completion 2011-10-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (phase I) | 3 years
  Dose-limiting toxicity (phase I)
Maximum-tolerated dose (phase I) | 3 years
  Maximum-tolerated dose (phase I)
Freedom from progression for 3 years (phase II) | 3 years
  Freedom from progression for 3 years (phase II)

SECONDARY OUTCOMES:
Time to biochemical, local and distant failure (phase II) | 3 years
  Time to biochemical, local and distant failure (phase II)
Disease-specific survival (phase II) | 3 years
  Disease-specific survival (phase II)
Overall survival rate (phase II) | 3 years
  Overall survival rate (phase II)
Adverse events as assessed by NCI CTCAE v. 4.0 | 3 years
  Adverse events as assessed by NCI CTCAE v. 4.0

CONTACTS AND LOCATIONS:
Overall Officials: David A. Pistenmaa, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States